CLINICAL TRIAL: NCT04541342
Title: Second-look Arthroscopic Evaluation of Cartilage Regeneration After Medial Opening-wedge High Tibial Osteotomy
Brief Title: Arthroscopic Evaluation of Cartilage Regeneration After Opening-wedge High Tibial Osteotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Sayed Mohamed, physician, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: arthroscopy with HTO
Record Dates: First submitted 2020-08-28; First posted 2020-09-09 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Intervention Model Description: quasi experimental one group pretest posttest study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- osteoarthritic with genu varus (Experimental): initial arthroscopy and high tibial osteotomy to be followed later by a second look arthroscopy with plate removal
  Interventions: Procedure: initial arthroscopy with medial opening-wedge high tibial osteotomy fixed by a plate system then second look arthroscopy with plate removal

INTERVENTIONS:
Procedure: initial arthroscopy with medial opening-wedge high tibial osteotomy fixed by a plate system then second look arthroscopy with plate removal — It is a joint preserving procedure especially preferred in young patients for whom arthroplasty is not desirable. The procedure promotes regeneration by causing lateral shift of the weight-bearing axis, thus decreasing load on the medial compartment and widening the medial joint space.Many of the patients complains of irritation through the plate and wish metal removal after healing of the osteotomy.All patients will undergo initial arthroscopy before high tibial osteotomy (HTO). During arthroscopy, debridement of the degenerate tissues and meniscal tears if present will be performed. Then opening-wedge high tibial osteotomy (OWHTO) will be performed and fixed by a plate system. Second-look arthroscopy will be conducted at the time of plate removal after healing of the osteotomy. This will be after about 6 months up to one year.

SUMMARY:
Osteoarthritis of the knee is a common problem causing significant knee pain and disability. Medial compartment osteoarthritis is predisposed to by varus deformity of the knee. High tibial osteotomy is a well-established method for treatment of medial unicompartmental knee osteoarthritis and correction of varus deformity.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative joint disease characterized by erosion of the articular cartilage, hypertrophy of the bone at the margins and subchondral sclerosis. Osteoarthritis of the knee is a common problem causing significant knee pain and disability. Medial compartment osteoarthritis is predisposed to by varus deformity of the knee. High tibial osteotomy is a well-established method for treatment of medial unicompartmental knee osteoarthritis and correction of varus deformity. It is a joint preserving procedure especially preferred in young patients for whom arthroplasty is not desirable. The procedure promotes regeneration by causing lateral shift of the weight-bearing axis, thus decreasing load on the medial compartment and widening the medial joint space. The methods for اigh tibial osteotomy include opening-wedge osteotomy and closed wedge osteotomy. An opening-wedge osteotomy has become increasingly popular compared to the other technique. One of the disadvantages of this technique is that the plate is placed subcutaneously on the medial aspect of the proximal tibia. Many of the patients complains of irritation through the plate and wish metal removal after healing of the osteotomy. Few papers assessed regeneration of the articular cartilage after medial opening-wedge osteotomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age younger than 65 years
2. Medial joint line tenderness
3. BMI less than 30
4. Varus tibiofemoral malalignment
5. Range of motion in the knee joint maintained from greater than 100 degrees of flexion to less than 15 degrees of flexion contracture
6. Osteoarthritis of the knee with any degree of cartilage damage provided that the cartilage damage in the lateral compartment not exceeding Outerbridge grade 2
7. No associated ligamentous functional instability

Exclusion Criteria:

1. Age older than 65 years
2. Severe Lateral compartment osteoarthritis (Outerbridge grade 3 or 4)
3. Flexion contracture of greater than 15 degrees
4. Inflammatory arthritis, post-traumatic osteoarthritis, active knee infection

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Arthroscopic assessment of cartilage regeneration after high tibial osteotomy | 6 months after high tibial osteotomy
  By use of Outerbridge classification of chondral lesions during arthroscopy, comparison will be made between cartilage status before and after high tibial osteotomy according to the Outerbrigde classification which classifies cartilage lesions into grades of 0 through IV. Grade 0 signifies normal cartilage.
  Grade I chondral lesions are characterized by softening and swelling, which often require tactile feedback with a probe or other instrument to assess. Grade II lesion describes a partial-thickness defect with fissures that do not exceed 0.5 inches in diameter or reach subchondral bone.
  Grade III is fissuring of the cartilage with a diameter > 0.5 inches with an area reaching subchondral bone.
  The most severe is Grade IV, which includes erosion of the articular cartilage that exposes subchondral bone.

SECONDARY OUTCOMES:
Post-operative limb alignment | 6 months after high tibial osteotomy
  by use of bilateral standing anteroposterior full-length views of both lower limbs before high tibial osteotomy and at time of plate removal. The tibiofemoral angle will be measured to detect the degree of varus correction.

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Assiut University Hospitals, Asyut
  - AssiutU Hospitals, Asyut

REFERENCES:
- [Background] Kim KI, Seo MC, Song SJ, Bae DK, Kim DH, Lee SH. Change of Chondral Lesions and Predictive Factors After Medial Open-Wedge High Tibial Osteotomy With a Locked Plate System. Am J Sports Med. 2017 Jun;45(7):1615-1621. doi: 10.1177/0363546517694864. Epub 2017 Mar 14. PMID 28291955
- [Background] Slattery C, Kweon CY. Classifications in Brief: Outerbridge Classification of Chondral Lesions. Clin Orthop Relat Res. 2018 Oct;476(10):2101-2104. doi: 10.1007/s11999.0000000000000255. No abstract available. PMID 29533246
- [Background] Koshino T, Wada S, Ara Y, Saito T. Regeneration of degenerated articular cartilage after high tibial valgus osteotomy for medial compartmental osteoarthritis of the knee. Knee. 2003 Sep;10(3):229-36. doi: 10.1016/s0968-0160(03)00005-x. PMID 12893144
- [Derived] AbdelKawi AF, El-Assal MA, Abdelhamid MM, Sayed AM. Arthroscopic evidence of improvement in cartilage lesions after medial opening-wedge high-tibial osteotomy with valgus correction and its positive impact on clinical outcomes, a prospective study. Int Orthop. 2025 Aug;49(8):1879-1885. doi: 10.1007/s00264-025-06552-x. Epub 2025 Jun 2. PMID 40455268